CLINICAL TRIAL: NCT00025558
Title: Dose Escalation of Temozolomide in Combination With Thiotepa and Carboplatin With Autologous Stem Cell Rescue in Patients With Malignant Brain Tumors With Minimal Residual Disease
Brief Title: Combination Chemotherapy Followed by Peripheral Stem Cell Transplantation or Bone Marrow Transplantation in Treating Patients With Brain Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068973; P30CA016087 (NIH); NYU-0006H; NCI-G01-2022
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood central nervous system germ cell tumor; recurrent adult brain tumor; adult medulloblastoma; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult central nervous system germ cell tumor; adult pineoblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood medulloblastoma; recurrent childhood ependymoma; adult giant cell glioblastoma; adult gliosarcoma; adult anaplastic ependymoma; adult supratentorial primitive neuroectodermal tumor (PNET)
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Medulloblastoma; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Pinealoma; Familial ependymoma; Gliosarcoma; Ependymoma | interventions — Filgrastim; Carboplatin; Temozolomide; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: temozolomide
Drug: thiotepa
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation or bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining temozolomide, thiotepa, and carboplatin followed by peripheral stem cell transplantation or bone marrow transplantation in treating patients who have brain cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of temozolomide in combination with thiotepa and carboplatin followed by autologous peripheral blood stem cell or bone marrow transplantation in patients with recurrent high-grade brain tumors with minimal residual disease or newly-diagnosed malignant glioma with minimal residual disease following irradiation.

OUTLINE: This is a dose-escalation study of temozolomide.

Patients receive filgrastim (G-CSF) subcutaneously (SC) once daily for 3 consecutive days. After the third dose of G-CSF, patients undergo leukapheresis to collect peripheral blood stem cells (PBSC). Patients who do not have adequate PBSC may undergo bone marrow harvest.

Patients then receive oral temozolomide every 12 hours on days -10 to -6 and thiotepa IV over 3 hours and carboplatin IV over 4 hours on days -5 to -3.

PBSC or bone marrow are reinfused on day 0. Beginning on day 1, patients receive G-CSF SC or IV until blood counts recover.

Cohorts of 3-6 patients receive escalating doses of temozolomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at day 42, at 3 months, every 3 months for 2 years, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 18-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following malignant brain tumors:

  * Anaplastic astrocytoma
  * Glioblastoma multiforme
  * Anaplastic oligodendroglioma
  * Medulloblastoma
  * High-grade ependymoma
  * Germ cell tumors
  * Pineoblastoma
  * Other primitive neuroectodermal tumors
* Recurrent disease or resistant to conventional therapy (e.g., surgery, radiotherapy, or standard chemotherapy)

  * No prior myeloablative doses of thiotepa OR
* Newly diagnosed malignant glioma with minimal residual disease after prior radiotherapy

  * Minimal residual disease is defined as tumor with maximum diameter of less than 1.5 cm by MRI and no corticosteroid dependency

PATIENT CHARACTERISTICS:

Age:

* Over 1 to under 50

Performance status:

* Karnofsky 70-100% OR
* Lansky 70-100%

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 10 g/dL (transfusion allowed)

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT/SGPT less than 2.5 times ULN
* Alkaline phosphatase less than 2.5 times ULN

Renal:

* Creatinine less than 1.5 times ULN
* Creatinine clearance at least 70 mL/min
* BUN less than 1.5 times ULN

Cardiovascular:

* Ejection fraction greater than 50% OR
* Shortening fraction greater than 27%
* No evidence of myocardial ischemia on EKG if over 40 years of age

Other:

* HIV negative
* No AIDS-related illness
* No frequent vomiting or medical condition that would preclude oral medication (e.g., partial bowel obstruction)
* No other malignancy within the past 2 years except surgically cured carcinoma in situ of the cervix or basal cell or squamous cell skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 2 weeks since prior biologic therapy or immunotherapy

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics
* At least 6 weeks since prior radiotherapy and recovered
* At least 6 weeks since prior brachytherapy or radiosurgery

Surgery:

* See Disease Characteristics
* Recovered from prior major surgery

Ages: 1 Year to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-10; Primary Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L. Gardner, MD, Study Chair — NYU Langone Health
Locations (4):
- United States (3):
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia